CLINICAL TRIAL: NCT05821283
Title: Does Physical Activity Provide Additional Benefit In Patients With Rotator Cuff Related Shoulder Pain? A Randomized Controlled Trial
Brief Title: Does Physical Activity Provide Additional Benefit In Patients With Rotator Cuff Related Shoulder Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Derya Celik, Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR2023
Record Dates: First submitted 2023-03-16; First posted 2023-04-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Rotator Cuff Injuries
Keywords: rotator cuff; physical activity; shoulder pain
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity; Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Group (Experimental): The Physical Activity (PAG) was included in an exercise program consisting of supervised exercise and physical activity (30 minutes of moderate-intensity walking).
  Interventions: Procedure: exercise program consisting of supervised exercise and physical activity
- Control Group (Active Comparator): The Control Group (CG) was included in the program consisting of only supervised exercises.
  Interventions: Procedure: exercise program consisting of only supervised exercises.

INTERVENTIONS:
Procedure: exercise program consisting of supervised exercise and physical activity — The Physical Activity Group (PAG) included in an exercise program consisting of supervised exercise and physical activity (30 minutes of moderate-intensity walking). Patients received 6 week (2-3 times a week) rehabilitation program composed of 15 physical therapy sessions.The physical activity program was applied as moderate intensity (maximum heart rate 50-70%) walking exercise. The patients were recommended to walk for 30 minutes, 3 days a week (total of 90 minutes) for the first 3 weeks, and 30 minutes 5 days a week (total of 150 minutes) for the 2nd 3 weeks
  Arms: Physical Activity Group
Procedure: exercise program consisting of only supervised exercises. — The Control Group (CG) included in the program consisting of only supervised exercises. Patients received 6 week (2-3 times a week) rehabilitation program composed of 15 physical therapy sessions
  Arms: Control Group

SUMMARY:
Rotator cuff-related shoulder pain (RCRSP) are among the most common musculoskeletal disorders and can be associated with pain, weakness, shoulder dysfunction and kinesiophobia. The management could be surgery or nonsurgical options such as medical treatment, education, activity modifications and physiotherapy. Physical activity is defined as any body movement produced by skeletal muscles that requires a certain amount of energy expenditure. Regular physical activity is proven to help prevent and manage many diseases. Beyond these people, doing physical activity have better mental health, emotional wellbeing, quality of life and lower rates of mental illness. Additionally, physical activity and exercise applications are used as an alternative method to reduce the severity and frequency of pain in patients with chronic pain. Investigators reviewed the literature, we could not find any randomized controlled trial on the effectiveness of physical activity in studies conducted with patients with RCRSP. Investigators hypothesized that adding physical activity to the treatment of RCRSP would make a significant difference. Therefore, the aim of this study was to investigate the effect of physical activity applied in addition to supervised exercise on pain, functional status and quality of life in patients with RCRSP.

DETAILED DESCRIPTION:
Rotator cuff-related shoulder pain (RCRSP) are among the most common musculoskeletal disorders and can be associated with pain, weakness, shoulder dysfunction and kinesiophobia. The management could be surgery or nonsurgical options such as medical treatment, education, activity modifications and physiotherapy. However, none of this interventions was found best additionally 30% of individuals do not report significant improvement. Physical activity is defined as any body movement produced by skeletal muscles that requires a certain amount of energy expenditure. Regular physical activity is proven to help prevent and manage many diseases such as heart disease, stroke, several cancers, diabetes, hypertension and obesity. Beyond these people, doing physical activity have better mental health, emotional wellbeing, quality of life and lower rates of mental illness. Additionally, physical activity and exercise applications are used as an alternative method to reduce the severity and frequency of pain in patients with chronic pain.

Physical activity is defined as any body movement produced by skeletal muscles that requires a certain amount of energy expenditure. Investigators reviewed the literature, investigators could not find any randomized controlled trial on the effectiveness of physical activity in studies conducted with patients with RCRSP. Investigators hypothesized that adding physical activity to the treatment of RCRSP would make a significant difference. Therefore, the aim of this study was to investigate the effect of physical activity applied in addition to supervised exercise on pain, functional status and quality of life in patients with RCRSP. This study was prospective, randomized controlled; assessor-blinded trial was performed to compare the effectiveness of physical activity in addition to supervised exercise in patients with RCRSP. According to the power analysis result, 46 patients were randomized into two groups(Treatment Group=23, Control Group=23).The Physical Activity Group (PAG) was included in an exercise program consisting of supervised exercise and physical activity (30 minutes of moderate-intensity walking). The Control Group (CG) was included in the program consisting of supervised exercises only. The treatment lasted for a total of 6 weeks. The primary outcome was Numeric Pain Rating Scale (NPRS)-activity and secondary outcomes were Numeric Pain Rating Scale (NPRS)-night The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment (ASES), Quick Disabilities of The Arm, Shoulder and Hand Questionnaire (Quick DASH), Rotator Cuff Quality of Life (RC-QOL) Western-Ontario Rotator Cuff Index (WORC) and Global Rate of Changes (GRC) scores.

ELIGIBILITY:
Inclusion Criteria:

* Subject age of more than 40 years
* Having at least 3 months of unilateral shoulder pain
* Presence of painful arc
* Positive Hawkins Kennedy test or positive Neer sign
* Painful shoulder abduction and external rotation with resistance
* Absence of radiological findings of fracture in the humeral greater tubercle or glenoid cavity
* Obtaining informed written consent

Exclusion Criteria:

* Having a massive rotator cuff tear (confirmed with Magnetic Resonance (MR) and positive lag sign)
* History of trauma related to onset of symptoms
* Having undergone surgery on the same shoulder
* Frozen shoulder
* Symptomatic cervical spine pathology
* Shoulder instability
* Presence of shoulder problems caused by systemic diseases, neurological disorders
* Having psychological, emotional or cognitive problems
* Previous shoulder surgery and steroid injections
* Engagement of regular physical activity

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS)-activity | change from baseline NPRS at 6 week
  The pain will be measured at activity using a NPRS. Patients are asked to rate their pain ranging from 0 to 10 (0: no pain, 10: the worst pain imaginable)

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS)-night | change from baseline NPRS at 6 week
  The pain will be measured at night using a NPRS. Patients are asked to rate their pain ranging from 0 to 10 (0: no pain, 10: the worst pain imaginable)
The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment (ASES) | change from baseline ASES score at 6 week
  The ASES score ranges from 0-100. Higher scores indicate better functional ability.
Quick Disabilities of The Arm, Shoulder and Hand Questionnaire (Quick DASH) | change from baseline Quick DASH score at 6 week
  The Quick DASH is a 11-item questionnaire used to assess upper limb functionality. The score ranges from 0 (no disability) to 100 (most severe disability).
Rotator Cuff Quality of Life (RC-QOL) | change from baseline RC-QOL score at 6 week
  RC-QOL consists of 34 items and each question consists of a line between 0 and 100. The point on the line is measured with a ruler and the value is written. Higher values indicate better quality of life.The total score ranges from 0 to 3400, with higher scores indicating higher quality of life. The percentage (%) score can also be calculated by dividing the total score obtained by 34.
Western-Ontario Rotator Cuff Index (WORC) | change from baseline WORC score at 6 week
  WORC-Emotions consist of 3 items. Each question is answered with a 100 mm Visual Analog Scale (VAS). Lower scores indicate better quality of life motions consist of 3 items. Each question is answered with a 100 mm Visual Analog Scale (VAS). Lower scores indicate better quality of life.The total score ranges from 0 to 300, with lower scores indicating higher quality of life. The percentage (%) score can also be calculated by dividing the total score obtained by 3.
Global Rate of Changes (GRC) | change from baseline GRC score at 6 week
  GRC is used to determine the effectiveness of treatment by questioning the patient's improvement or worsening over time. In our study, a 7-point scale (-3: much worse, -2: worse, -1: slightly worse, 0: same, 1: slightly better, 2: quite good, 3: much better) was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes